CLINICAL TRIAL: NCT04231708
Title: Effects of Pharmacological Stress and Repetitive Transcranial Magnetic Stimulation Interventions on Executive Function in Opioid Use Disorder
Brief Title: Effects of Pharmacological Stress and rTMS on Executive Function in Opioid Use Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Principal Investigator, Wayne State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DL-STR-OUD
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Yohimbine; Hydrocortisone

STUDY DESIGN:
Intervention Model Description: Double-blind, 10Hz left dlPFC rTMS (vs. sham) X pharmacological stressor (vs. placebo) within-subject, randomized crossover design.
Who Masked: Participant, Outcomes Assessor
Masking Description: Placebo (lactose) for pharmacological stressor, and sham for dlPFC rTMS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- placebo stressor, sham rTMS (Placebo Comparator): Placebo stressor (lactose) + sham (inactive) rTMS over the left dlPFC
  Interventions: Drug: Placebo; Device: Sham rTMS
- placebo stressor, active rTMS (Experimental): Placebo stressor (lactose) + active 10Hz rTMS over the left dlPFC
  Interventions: Device: Active rTMS; Drug: Placebo
- active stressor, sham rTMS (Experimental): Stressor (yohimbine 54mg + hydrocortisone 20mg) + sham (inactive) rTMS over the left dlPFC
  Interventions: Drug: Yohimbine + Hydrocortisone; Device: Sham rTMS
- active stressor, active rTMS (Experimental): Stressor (yohimbine 54mg + hydrocortisone 20mg) + active 10Hz rTMS over the left dlPFC
  Interventions: Drug: Yohimbine + Hydrocortisone; Device: Active rTMS

INTERVENTIONS:
Drug: Yohimbine + Hydrocortisone — Yohimbine (54mg bulk powder inside capsule) administered in combination with Hydrocortisone (20mg tablet inside capsule)
  Arms: active stressor, active rTMS; active stressor, sham rTMS
Device: Active rTMS — 10Hz rTMS over the left dlPFC
  Arms: active stressor, active rTMS; placebo stressor, active rTMS
Drug: Placebo — lactose (inside capsule)
  Arms: placebo stressor, active rTMS; placebo stressor, sham rTMS
Device: Sham rTMS — inactive stimulation over the left dlPFC
  Arms: active stressor, sham rTMS; placebo stressor, sham rTMS

SUMMARY:
This preliminary study is designed to evaluate mechanisms by which excitatory dorsolateral prefrontal cortex (dlPFC) repetitive transcranial magnetic stimulation (rTMS) (vs. sham) and pharmacological stress (vs. placebo) alter behavior in non-treatment seeking individuals with opioid use disorder (OUD). Specific Aims are to (1) Evaluate how stress impacts domains of behavior including (1a) executive function and (1b) opioid-seeking behavior; and (2) Determine whether rTMS stimulation attenuates (2a) executive dysfunction, (2b) stress-reactivity, and (2c) opioid-seeking in individuals with OUD not receiving treatment.

DETAILED DESCRIPTION:
This study will use a double-blind, 10Hz left dlPFC rTMS (vs. sham) and pharmacological stressor ([yohimbine + hydrocortisone] vs. placebo) within-subject, randomized crossover design. Each participant will complete 4 sessions (stressor vs. placebo, crossed with rTMS vs. sham), each separated by at least 1 week. Participants will complete these 4 (2x2 within subject) test conditions in randomized order: sham rTMS/placebo stress, sham rTMS/active stress, active rTMS/ placebo stress, and active rTMS/active stress.

The PI will perform randomization using a Latin Square and will assign participants to conditions and prepare medication (stressor or placebo) for each participant's sessions. The PI will keep others blinded and will not be involved in study assessments.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-5 criteria for OUD;
* Age 21-60 yr;
* Right handed;
* Males and non-pregnant/non-lactating females;
* cognitively intact (total IQ score >80 on Shipley Institute of Living Scale);
* Screening cardiovascular indices within ranges for safe use of the pharmacological stressor: resting HR 50-90 bpm, systolic BP 90-140 mmHg, and diastolic BP 50-90 mmHg;
* Use alcohol and/or marijuana <3 times/week; each "time" should consist of <1 marijuana "joint" equivalent and <3 alcoholic drinks.

Exclusion Criteria:

* Under influence of any substance during session;
* Past 7-day use of illicit drugs other than opioids (except marijuana, which is legal in Michigan);
* Urinalysis positive for cocaine metabolites, benzodiazepines, barbiturates, amphetamines or pregnancy;
* Medical conditions prohibiting use of rTMS (e.g. seizure history; based on rTMS screening questionnaire);
* Lifetime diagnosis of: psychotic disorder, bipolar disorder, generalized anxiety disorder, or obsessive compulsive disorder; major depression in the past 5 years; or potentially antisocial personality disorder (if the clinical psychologist judges such behaviors to be potentially disruptive or unsafe in our lab);
* Past-year SUD other than OUD;
* Acute/unstable illness: conditions making it unsafe for participation (e.g. neurological, cardiovascular, pulmonary, or systemic diseases);
* Lactose intolerance (placebo dose);
* Any prohibited medications: medications that lower seizure threshold, psychiatric medications, prescription pain medications, or blood pressure medications;
* Chronic head or neck pain; and
* Past-month participation in a research study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Color-Word Stroop Task | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  measures cognitive control in response to opioid-related words.
Digit Span Task | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  measures verbal working memory. Participants are asked to repeat strings of numbers of increasing length, both forward and backward.
Wisconsin Card Sorting Task | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  measures ability to shift set and assesses cognitive flexibility.
Emotion Regulation Task | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  subjects rate the unpleasantness and arousal of different emotional pictures
Positive and Negative Affect Schedule | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  subjects rate their positive and negative affect
State-Trait Anxiety Inventory | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  subjects rate their level state anxiety
Monetary Incentive Delay Task | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  Participants respond to a visual target that follows 2 different cues: incentive or non-incentive. No reward or punishment occurs on non-incentive trials. On incentive trials, participants must respond within a fixed amount of time. In the reward condition, responses within that time result in receiving the incentive , else nothing. In the punishment condition, the participant will lose money if they do not respond within the time limit
Delay Discounting Task | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  Participants perform a brief (<1min) hypothetical version of the traditional monetary task with a 5-trial adjusting delay previously validated to rapidly assess discount rate
Drug/Money Choice Task | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  participants choose hypothetically between a constant amount of their preferred opioid ($10 unit dose) or money ($2)
Systolic blood pressure | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  millimeters mercury (mmHg)
Diastolic blood pressure | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  millimeters mercury (mmHg)
Heart rate | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  beats per minute
Saliva cortisol level | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  measure of the activity of the HPA axis
Saliva alpha-amylase level | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  indirect measure of adrenergic stimulation
Serum prolactin level | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  indirect measure of dopamine stimulation
Serum brain derived neurotrophic factor (BDNF) level | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  indirect measure of brain derived neurotrophic factor activation
Relative electroencephalogram (EEG) gamma power | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  Prefrontal gamma (25-100 Hz) EEG power, relative to slow-wave EEG power, is a stress biomarker

SECONDARY OUTCOMES:
Opioid craving | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  Desire for Drug Questionnaire total score; higher scores indicate greater craving
Opioid agonist symptoms | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  Opiate-32 questionnaire agonist symptom total score; higher scores indicate greater opioid symptom severity
Opioid withdrawal symptoms | change from pre- to post-intervention in each of 4 sessions (through study completion, about 1 month total)
  Opiate-32 questionnaire withdrawal symptom total score; higher scores indicate greater withdrawal severity

CONTACTS AND LOCATIONS:
Locations (1):
- Tolan Park Medical Building, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No